CLINICAL TRIAL: NCT07352332
Title: A Prospective Observational Study of Immune Profiling in Childhood-Onset Systemic Lupus Erythematosus Under CD3×CD19 Bispecific T-Cell Engager Exposure
Brief Title: Immune Profiling of Refractory cSLE Exposed to CD3×CD19 BiTE
Acronym: BiTE-cSLE-IP
Status: Recruiting | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhang Xiaojing, MD, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: ZhangXJ1984
Record Dates: First submitted 2025-12-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Childhood-onset Systemic Lupus Erythematosus
Keywords: Childhood-onset Systemic Lupus Erythematosus; Refractory Systemic Lupus Erythematosus; Immune Profiling; Bispecific T-Cell Engager; Single-Cell Sequencing; Flow Cytometry
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CD3×CD19BiTE-Treated cSLE Cohort: This cohort includes pediatric patients with refractory SLE who are receiving CD3×CD19 BiTE therapy as part of routine clinical care. The study does not assign treatment; BiTE administration follows standard clinical decision-making. Participants will undergo longitudinal peripheral blood collection for immune profiling using flow cytometry and single-cell sequencing methods. Clinical data will be collected in parallel to explore associations between immune features and disease activity.

SUMMARY:
This prospective observational study aims to characterize the peripheral immune landscape of pediatric patients with childhood-onset systemic lupus erythematosus ( cSLE) who are receiving CD3×CD19 bispecific T-cell engager (BiTE) therapy under a separate, approved exploratory clinical study. The present study does not assign, modify, or influence any therapeutic interventions.

Peripheral blood samples are collected longitudinally at predefined time points in parallel with routine clinical follow-up. Immune profiling is performed using multiparameter flow cytometry, with single-cell sequencing conducted in a subset of samples to further explore cellular and molecular features. Clinical data, including disease activity indices and relevant serological biomarkers, are recorded concurrently.

The objective of this study is to describe immune cell dynamics and immune features associated with changes in disease activity in cSLE, and to explore potential biomarker candidates that may inform future immune-monitoring strategies and mechanistic research in this population.

DETAILED DESCRIPTION:
Childhood-onset systemic lupus erythematosus (cSLE) is a severe autoimmune disease characterized by early disease onset, frequent multi-organ involvement, high disease activity, and a relapsing-remitting clinical course. Despite treatment with conventional immunosuppressive agents and biologic therapies, a subset of pediatric patients continues to experience refractory or persistently active disease.

CD3×CD19 bispecific T-cell engagers (BiTEs) redirect endogenous T cells to eliminate CD19-positive B cells and have demonstrated potent immunologic effects in B-cell malignancies. In cSLE, CD3×CD19 BiTE therapy has been administered in a limited number of patients under a separate, approved exploratory clinical study, where preliminary clinical observations suggested immune changes accompanied by improvement in disease activity. However, the immunologic effects and immune dynamics associated with CD3×CD19 BiTE exposure in cSLE have not been systematically characterized, and longitudinal immune profiling data in this context remain scarce.

The present study is designed as a prospective, observational, single-center cohort study. It does not assign, modify, or influence any therapeutic interventions. All participants receive CD3×CD19 BiTE therapy solely as part of an independent exploratory clinical protocol, and the current study focuses exclusively on immune profiling under this predefined treatment background.

Peripheral blood samples are collected longitudinally at predefined time points before and after CD3×CD19 BiTE exposure, in parallel with routine clinical follow-up. Immune profiling is primarily performed using multiparameter flow cytometry to quantify the proportions, phenotypes, and activation states of major immune cell populations, including B-cell and T-cell subsets. In a subset of samples, single-cell sequencing is conducted to further explore cellular heterogeneity, transcriptional features, and potential immune pathways associated with observed immune changes.

Clinical data are collected concurrently, including disease activity indices (such as SLEDAI), serological markers (e.g., complement levels and anti-double-stranded DNA antibodies), and organ-related clinical parameters reflecting multi-organ involvement. These clinical variables are integrated with immune profiling data to explore associations between immune features and changes in disease activity.

The primary aim of this study is to describe the peripheral immune landscape and immune cell dynamics in patients with cSLE exposed to CD3×CD19 BiTE therapy. Secondary objectives include exploring immune features associated with changes in disease activity and identifying candidate immunologic biomarkers that may inform future immune-monitoring strategies or mechanistic studies. This study does not evaluate the efficacy or safety of CD3×CD19 BiTE therapy.

By systematically integrating longitudinal immune profiling with clinical data, this observational study seeks to provide foundational immunologic insights into cSLE under CD3×CD19 BiTE exposure and to support future hypothesis-driven research in immune monitoring and personalized immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria:

  1. Age ≥ 5 years.
  2. Diagnosis of systemic lupus erythematosus (SLE) confirmed according to the 2019 EULAR/ACR classification criteria.
  3. Refractory or persistently active SLE, defined by clinical evaluation and meeting at least one of the following conditions:

  <!-- -->

  1. Inadequate response to prior standard treatments, including oral glucocorticoids, antimalarial agents, conventional immunosuppressants (cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, cyclosporine, tacrolimus, sirolimus, leflunomide), and biologic therapies (telitacicept, belimumab, rituximab).
  2. Moderate to high disease activity, such as a SLEDAI score ≥ 6. 4.Receiving CD3×CD19 bispecific T-cell engager (BiTE) therapy as part of routine clinical management, with traceable dosing information and treatment timeline.

  5.Availability of peripheral blood samples collected before and/or after CD3×CD19 BiTE exposure, obtained during routine clinical assessment or prospective follow-up, that are suitable for immunologic analyses.

  6.Prior informed consent obtained in a related clinical study or clinical care context that explicitly permits the storage and secondary use of biological samples and associated clinical data for disease-related scientific research, including prospective analyses during subsequent follow-up; and willingness of the child to cooperate with study follow-up procedures, as appropriate.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded:

1. Inability to obtain peripheral blood samples of adequate quality for immunologic analyses, including insufficient sample volume, severe hemolysis, or failure to meet predefined cell viability criteria.
2. Presence of acute severe infection, acute organ decompensation, or other acute medical conditions that may substantially interfere with immune profiling analyses.
3. Significant risk associated with blood sampling, such as severe anemia, serious coagulation disorders, or other conditions deemed by the investigator to pose unacceptable risk for phlebotomy.
4. Inability to obtain essential clinical data required for immune-clinical correlation analyses (e.g., disease activity scores, complement levels, autoantibody results, or renal parameters).
5. Refusal of the legal guardian to allow participation or withdrawal of permission for use of biological samples, or lack of assent from the child when applicable.
6. Any other condition that, in the opinion of the investigator, may compromise study completion, data integrity, or participant safety.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients with childhood-onset systemic lupus erythematosus (cSLE) who have refractory or persistently active disease and are receiving CD3×CD19 BiTE therapy under a separate, approved exploratory clinical study. Participants are enrolled in this prospective observational cohort for longitudinal immune profiling using peripheral blood samples, without assignment or modification of therapeutic interventions.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in proportions and phenotypic characteristics of peripheral blood immune cell subsets | From baseline through 52 weeks
  Quantitatively characterize longitudinal changes in the proportions, phenotypes, and activation status of major peripheral immune cell populations (including B cells, T cells, and other relevant subsets) assessed by immunologic assays (primarily multiparameter flow cytometry; single-cell profiling may be used when available) in pediatric patients with refractory SLE treated with CD3×CD19 BiTE.

SECONDARY OUTCOMES:
Association between changes in peripheral blood immune cell subsets and disease activity indices | From baseline through 52 weeks
  Assessment of associations between longitudinal changes in peripheral blood immune cell subsets (cell subset proportions and/or phenotypic/activation markers) and disease activity indices during follow-up after CD3×CD19 BiTE exposure.
Single-cell sequencing-derived gene expression and pathway activity profiles in peripheral blood immune cells | From baseline through 12 weeks
  In selected samples, assessment of single-cell sequencing-derived molecular profiles, including differentially expressed genes, pathway activity, and inferred cell-cell communication signals in peripheral blood immune cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No